CLINICAL TRIAL: NCT03978026
Title: Evaluation de l'efficacité Sur la Vigilance et Les Performances de Conduite simulée d'Une Sieste effectuée Dans Des Environnements différents, Dont le Module SOMBOX
Brief Title: Vigilance and Simulated Driving After a Nap
Acronym: SOMBOX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Basic Science
Other Study IDs: ID RCB 2018-A02253-52
Record Dates: First submitted 2019-02-25; First posted 2019-06-06 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2019-02

CONDITIONS: Healthy Volunteers
Keywords: Nap; vigilance; cognition; driving simulation

STUDY DESIGN:
Intervention Model Description: Participant is evaluated in 4 situations :
  * nap in a bed
  * nap on a car sit
  * nap in the Sombox
  * no nap sitting on a car sit
Who Masked: Investigator
Masking Description: Participants will be recorded by technicians and results stored anonymously for traitement
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- nap in a bed (Experimental): the participants take a nap of 30 min in a bed in a bedroom
  Interventions: Behavioral: Nap
- nap in an armchair (Experimental): the participants take a nap of 30 min in a car sit in a bedroom
  Interventions: Behavioral: Nap
- nap in teh Sombox (Experimental): the participants take a nap of 30 min in the micro-hotel Sombox
  Interventions: Behavioral: Nap
- no nap in a bed (Sham Comparator): the participant stay awaked for 30 min in a bed in a bedroom
  Interventions: Behavioral: Nap

INTERVENTIONS:
Behavioral: Nap — Each participant is compared to himself in 4 conditions,

SUMMARY:
The objective of this study is to assess the effectiveness of naps under different environmental conditions and a rest without nap, on driving, alertness and psychomotor performance.

This study also aims to record during nap time, sleep, body temperature and heart rate.

DETAILED DESCRIPTION:
Nap time is one of the most effective means of combating decreased alertness throughout the day and maintaining cognitive and psychomotor performance.

As such, it is recommended for long-haul drivers driving their vehicle. However, these drivers have no alternative but to sleep in their seats. These conditions are not optimal for producing quality sleep. The motorcyclist, for his part, has no chance of sleeping without finding a place to feel safe to give himself up to sleep. On these bases, SOMBOX has developed a mini-hotel allowing drivers to find an optimized place to take a nap.

Investigators propose an experimental study to evaluate the effectiveness, on simulator driving performance and on the results obtained during cognitive and motor testing, of a nap taken under three different conditions. The effect of the nap will be assessed by comparison to a rest awake.

This study should include healthy volunteer participants.

ELIGIBILITY:
Inclusion Criteria:

* -Male and female participants, aged 20 to 50 years in good health, good sleepers (>8h on average), not being extreme chronotypes, without sleep disorders, healthy, unmedicated, not working in shift work, having been licensed for at least 2 years and driving a minimum of 5000 km per year
* The need for the collection of the signature of informed consent
* The need to be affiliated with the social security system
* The need to understand French

Exclusion Criteria:

* participant with a sleep disorder, even if not medicated
* participant with extreme morning or evening chronotype
* pregnancy
* ill or medicated participant

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
driving performances | baseline
  number of lateral deviations of the vehicule
sleepiness (vigilance) | baseline
  Psychomotor vigilance test (PVT)
fatigue (vigilance) | baseline
  Karolinska Sleepiness Scale (KSS),
motor coordination (vigilance) | baseline
  the angle of the steering wheel

SECONDARY OUTCOMES:
sleep | baseline
  (EEG : Fz, Cz, F4-M1, C4-M1, O2-M1, F3-M2 et O1-M2),
temperature | baseline
  measured each minute with e-tact medical device
heart rate | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Gauthier, Study Chair — UMR 1075 COMETE
Locations (1):
- PFRS, Caen, France

IPD SHARING:
Plan to Share IPD: No